CLINICAL TRIAL: NCT01464593
Title: Phase II Open Label Trial of Thermal Ablation and Lyso-Thermosensitive Liposomal Doxorubicin (Thermodox) for Metastatic Colorectal Cancer (mCRC) Liver Lesions
Brief Title: Phase 2 Study of Thermodox as Adjuvant Therapy With Thermal Ablation (RFA) in Treatment of Metastatic Colorectal Cancer(mCRC)
Acronym: ABLATE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: trial design contingent on RFA optimization
Sponsor: Imunon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104-10-201
Record Dates: First submitted 2011-11-01; First posted 2011-11-03 (Estimated); Results first posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-09

CONDITIONS: Colon Cancer Liver Metastasis
Keywords: Colorectal Liver Metastasis; Colon Cancer; Liver Cancer; Liver Metastasis; Liver metastases
MeSH Terms: conditions — Colonic Neoplasms; Liver Neoplasms | interventions — liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thermodox (Experimental): Thermodox 50 mg/m2 intravenous infusion over 30 minutes starting 15 minutes before thermal ablation.
  Interventions: Drug: Lyso-Thermosensitive Liposomal Doxorubicin; Other: 5% Dextrose Solution; Drug: ThermoDox

INTERVENTIONS:
Drug: Lyso-Thermosensitive Liposomal Doxorubicin — Thermally sensitive liposomal doxorubicin 50 mg/m2 single 30 minute intravenous infusion.
  Other Names: Liposomal doxorubicin; Doxorubicin; Thermodox
Other: 5% Dextrose Solution — Single 30 minute intravenous infusion
Drug: ThermoDox — ThermoDox is a Lyso-thermosensitive Liposomal Doxorubicin designed to be used in conjunction with thermal ablation.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Thermodox, a thermally sensitive liposomal doxorubicin, in combination with thermal ablation in the treatment of hepatic colorectal liver metastases (CRLM).

DETAILED DESCRIPTION:
This is an open label phase II trial to evaluate the safety, feasibility, and efficacy of ThermoDox in combination wtih thermal ablation for the regional hepatic treatment of mCRC liver lesions.

Eligible colorectal cancer patients will unresectable liver metastases and be candidate for either radiofrequency ablation (RFA) or microwave ablation (MWA). All unresectable lesions must be targeted for ablation in in nor more than 2 thermal ablation/ThermoDox procedures.

Approximately 24 hours prior to treatment with ThermoDox, patients will start a regimen of prophylaxis (detailed in the Study Drug section below) against immediate hypersensitivity reactions.

Treatment will begin with a 50 mg/m2 ThermoDox infusion administered intravenously (IV) over 30 minutes. Thermal Ablation will be initiated a minimum of 15 minutes after start of the infusion and should be completed no later than 3 hours after starting the infusion. Subjects will have follow up visits on Day 14 and at months 1, 4, 7, 10,13, 16, 19, 22, and 25 (+ 7 days) or until study discontinuation.

At baseline and at each post-treatment clinic visit, patients will self-report their "quality of life" (QoL) using the 8-item FACT-Hepatobiliary Symptom Index (FHSI-8).

Contrast CT imaging studies or Magnetic Resonance Imaging (MRI)will be used to assess the effectiveness of therapy. CT or MRI scans will be obtained at baseline and at months 1, 4, 7, 10, 13, 16, 19, 22, and 25(+ 7 days)until local recurrence is seen, the subject has discontinued, or 2 years of follow-up have elapsed, whichever occurs first. All protocol-specified CT/MRI images will be centrally read by an independent radiology assessor.

Subjects will be followed for each efficacy endpoint local tumor control through 2 years after treatment. Secondary endpoints including Overall Survival, Time to Local Recurrence, PRO deterioration) will be evaluated until the event occurs, the subject is discontinued, or until 3 years following treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic diagnosis of colorectal cancer.
2. A minimum of 1 unresectable mCRC liver lesion at baseline clinically indicated for radiofrequency ablation (RFA) or microwave ablation (MWA).

   * Recurrent lesions may have been treated previously by resection or ablation.
   * Anticipated ablation volume will be no larger than either removal of 3 hepatic segments or removal of more than 30% of total liver volume (as per maximum surgical limit).
   * Patients may have resectable lesions that are treated surgically.
   * If additional lesions are discovered during the ablation treatment procedure that were undetectable at screening will be treated at the discretion of the physician and guided by local standard of care.
   * Confirm the lesions are malignant by a pretreatment biopsy or by a biopsy obtained during the ablation procedure.
3. Subjects with suspected or limited extra-hepatic mCRC are eligible provided thermal ablation is clinically indicated. Chemotherapy is not permitted within 5 half-lives or 30 days if shorter prior to initial study treatment through 30 days following final study treatment.
4. Male or female 18 years of age or older.
5. Are willing to sign an informed consent form.
6. Left Ventricular Ejection Fraction(LVEF) ≥ 50%
7. Willing to return to the study site for study visits.
8. Have ECOG performance status ≤ 2 and life expectancy of ≥ 6 months.

Exclusion Criteria:

1. Concomitant bowel surgery and/or synchronous colon resection.
2. Have serious illnesses including, but not limited to, congestive heart failure;life threatening cardiac arrhythmia; or myocardial infarction or cerebral vascular accident within the last 6 months.
3. Have previously received any doxorubicin (study subjects being considered for completion of treatment may have received ThermoDox previously).
4. Are pregnant or breast-feeding. In women of childbearing potential, a negative pregnancy test (serum) is required within 14 days prior to study treatment.
5. Women and men of childbearing potential who are not practicing an acceptable form of birth control (i.e. diaphragm, cervical cap, condom, surgical sterility or birth control pills.
6. Have any known allergic reactions to any of the drugs or liposomal components or intravenous imaging agents to be used in this study.
7. Have portal or hepatic vein tumor invasion/thrombosis.
8. Have INR > 1.5 times the institution's upper normal limit (UNL), except in subjects who are therapeutically anticoagulated for medical conditions unrelated to CRLM such as atrial fibrillation. Subjects may be re-screened after condition is treated or anticoagulant is withheld.
9. Have platelet count < 75,000/mm3, absolute neutrophil count < 1500/mm3, or Hgb < 10.0 g/dL (unless the hemoglobin value has been stable, the subject is cardiovascularly stable, asymptomatic, and judged able to withstand the RFA procedure).
10. Have serum creatinine ≥ 2.5 mg/dL or calculated creatinine clearance (CrCl) ≤ 25.0 mL/min.
11. Have serum bilirubin > 3.0 mg/dL.
12. Have serum albumin < 2.8 g/dL.
13. Have body temperature > 38.3°C immediately prior to study treatment.
14. Have contraindications to receiving doxorubicin HCl.
15. Are being treated with other investigational agents or use of an investigational agent within 5 half-lives or 30 days whichever is longer preceding the first dose of study medication.
16. Use of chemotherapy within 5 half-lives or 30 days, whichever is shorter, preceding the first dose of study medication and no chemotherapy planned for 30 days after ablation(s).
17. Have concurrent malignancy other than mCRC (subjects wtih treated squamous cell carcinoma of the skin or basal cell carcinoma of the skin maybe included) or ongoing medically significant active infection.
18. Documented HIV positive.
19. NYHA class III or IV functional classification for heart failure.
20. Evidence of hemochromatosis.
21. Have history of contrast induced nephropathy and unable to undergo MRI.
22. Have a history of Nephrogenic Systemic Fibrosis (NSF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Borys, M.D., Study Director — Imunon
Locations (4):
- United States (4):
  - UCLA, Los Angeles, California
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Hospital, Cleveland, Ohio
  - Rhode Island Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thermodox
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study terminated early due to lack of enrollment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Thermodox
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Determine the Local Tumor Control at 1 Year Post Randomization
Description: Subject's treated with thermal ablation in conjunction with Thermodox to evaluate local tumor control defined as complete ablation and does not experience recurrence within 1 cm of the ablation site.
Time Frame: 1 year
Population: Study terminated early due to lack of enrollment and data were not collected
Arm/Group | Thermodox
Number analyzed (Participants) | 0

2. Secondary Outcome: Evaluation of Safety
Description: Adverse events will be assessed through 1 month following study treatment(s). AE's after 1 month through the Month 25 assessment are reported if possibly, probably, or definitely related to study drug. Safety data will include physical exams, vital signs, ECGs, Echocardiograms/MUGA Scans, hematology, clinical chemistry and urinalysis.
Time Frame: 1 month
Population: Study terminated early due to lack of enrollment and data were not collected
Arm/Group | Thermodox
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Local Recurrence
Description: Measured as the time to local recurrence after ablation as measured from the date of randomization.
Time Frame: 2 years
Population: Study terminated early due to lack of enrollment and data were not collected
Arm/Group | Thermodox
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Description: Measured as time from randomization to death or the end of the study at month 37.
Time Frame: 3 years
Population: Study terminated early due to lack of enrollment and data were not collected
Arm/Group | Thermodox
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Thermodox
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No